CLINICAL TRIAL: NCT05576948
Title: Understanding the Early Natural History of Cerebral Palsy - A Prospective Cohort Study
Brief Title: Natural History of Cerebral Palsy Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cerebral Palsy Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0189
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with or at high risk of CP: Infants with a diagnosis of CP OR at high risk of CP as per the international Clinical Practice Guideline for early diagnosis of CP. In order to develop prognostic curves for motor function a minimum of 3 data points are required per participant. For this reason infants will be included if they are 12 months or younger (corrected age) at the time of enrolment.

SUMMARY:
The study will describe the natural history of cerebral palsy (CP) as children develop over the first 2 years of life.

DETAILED DESCRIPTION:
This study aims to describe the early natural history of cerebral palsy (CP) by mapping the development of infants with, or at-risk of CP, over the first two years of life. Infants will be assessed at regular intervals up to 24 months of age, across a variety of childhood development to provide the first comprehensive developmental trajectories of this group. In doing so, it will contribute to the existing knowledge of CP development to assist clinicians and therapists with accurate information on prognosis and provide targeted interventions early and at the 'just-right' challenge. Where indicated, individual participants' results from this study will be used to inform their therapy. This study is intended to form part of a larger multi-site international study.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be included if they have a diagnosis of CP or "at high risk of CP" and under the age of 12 months.
* Infants at high risk of CP as defined by any two (any combination) of the following:

  1. Neuroimaging predictive of a motor disability including the involvement of 1 or more of the following structures: sensori-motor cortex, Basal Ganglia, Posterior Limb of the Internal Capsule, pyramids.
  2. Trajectory of cramped synchronized general movements (GMs) on General Movement Assessment (GMA) OR absent fidgety GMs at fidgety age
  3. Hammersmith Infant Neurological Exam (HINE) scores <57 @ 3months or <60 @ 6months or <63 @9 months

     Infants will also be included if they meet BOTH of the following criteria (even if infants have a HINE score greater than the cut off scores stated above:

     i. Unilateral brain injury on neuroimaging (magnetic resonance imaging (MRI) or cranial ultrasound (CUS)) predictive of CP ii. Clinical signs of asymmetry

     Exclusion Criteria:
* Infants with progressive or neurodegenerative disorders or genetic disorders not associated with CP
* Infants with other disability diagnoses e.g. Down Syndrome

Ages: 3 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Infants with or at high-risk for CP
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Change in Motor skills | 3 months, 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Peabody: Gross and Fine motor skills
Change in Speech and Language skills | 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Bayley Scales of Infant and Toddler Development
Change in Cognitive skills | 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Bayley Scales of Infant and Toddler Development
Change in Neurologic assessment | 3 months, 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Hammersmith Infant Neurological Examination
Change in Musculoskeletal assessment | 3 months, 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Modified Tardieu Scale
Change in Musculoskeletal assessment | 9 months, 12 months, 18 months, 24 months (corrected age)
  Australian Spasticity Assessment Scale
Change in Musculoskeletal assessment | 18 months, 24 months corrected age
  Hip X-ray
Change in Vision | 6 months, 9 months, 12 months, 18 months, 24 months (corrected age)
  Previas
Vision | 3 months corrected age
  Ricci
Change in Sleep | 9 months, 12 months, 18 months, 24 months (corrected age)
  Sleep disturbances Scale for Children
Change in Feeding skills | 12 months, 18 months, 24 months (corrected age)
  Dysphagia Disorder Survey
Change in Self Care | 6 months, 12 months, 18 months, 24 months (corrected age)
  Pediatric Evaluation of Disability Inventory Computerized Assessment Test
Change in Adaptive Behavior | 12 months, 18 months, 24 months (corrected age)
  Infant Toddler Social Emotional Assessment
Change in Parent Well Being | 12 months, 18 months, 24 months (corrected age)
  Depression, Anxiety and Stress Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided